CLINICAL TRIAL: NCT06517706
Title: Brain Research and Integrative Neuroscience Network for COVID-19 (BRAINN)
Brief Title: Brain Research and Integrative Neuroscience Network for COVID-19
Acronym: BRAINN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cyprus (Other)
Responsible Party: Principal Investigator, Fofi Constantinidou, Professor of Psychology, University of Cyprus
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 101079001
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Training; Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Random Assignment
Who Masked: Participant, Care Provider
Masking Description: Participants will be randomly assigned to the experimental and control group. Both groups will receive cognitive rehabilitation. The experimental group control group will also active tDCS treatment whereas the control will receive inactive or sham tDCS treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Condition (Sham Comparator): Combination of cognitive training with sham tDCS
  Interventions: Behavioral: Categorization Program
- Experimental Condition (Experimental): Combination of cognitive training with active tDCS
  Interventions: Combination Product: Combination of tDCS (device) with cognitive training (behavioral)

INTERVENTIONS:
Combination Product: Combination of tDCS (device) with cognitive training (behavioral) — Participation in 15 one-hour sessions distributed over three weeks. During each session participants will receive two sessions of tDCS plus cognitive training with the Categorization Program
  Arms: Experimental Condition
Behavioral: Categorization Program — Participation in 15 one-hour sessions distributed over three weeks. During each session participants will receive cognitive training and sham tDCS
  Arms: Control Condition

SUMMARY:
The aim of the experimental study is to investigate two interventions for the management of cognitive symptoms resulting from long COVID. Participants will be randomly assigned into two interventions. 1. Categorization Program (CP) training with active tDCS or 2. Categorization Program training with sham tDCS.

DETAILED DESCRIPTION:
The two intervention protocols (digitalized CP and NIBS) required for this study have been developed and the required equipment (one existing and three new tDCS devices) has been acquired. Recruitment for the feasibility study is planned to begin in month 18, i.e., June 2024.

Changes in the design of the feasibility study have been made by the SC and in coordination with the Advisory Board. The changes were deemed necessary to improve the original study design to capture changes in cognition due to treatment. Specifically, the feasibility study will retain the two-group design (experimental and control). Forty participants with PCS will be recruited (instead of seventy, as originally planned). All participants will undergo the diagnostic protocols (the neuroimaging and neuropsychological assessments). Then, participants will be randomly assigned into two groups: the experimental, who will receive the active tDCS and CP intervention, and the control group, who will receive the sham tDCS and CP intervention. Following the intervention, all participants (experimental and control) will complete a series of dependent measures, including neuropsychological performance and quality of life measures. For neurophysiological measures, electroencephalography (EEG) has been replaced with functional near-infrared spectroscopy (fNIRS), which will be conducted both pre- and post-intervention. The current design will require a longer intervention period (as compared to the original design) and the complete delivery of the digitalized CP to maximize treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Reported cognitive difficulties due to COVID-19 infection
* WHO Long COVID criteria will be used

Exclusion Criteria:

* Significant history of neuropsychiatric conditions prior to contracting COVID-19; history of neurological conditions such as TBI, CVA, MS prior to contracting COVID-19.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Categorization Program Test 1 | Administered pre & post training with the Categorization Program, at 6 weeks
  Semantic knowledge and classification behavior
Categorization Program Test 2 | Administered pre & post training with the Categorization Program, at 6 weeks
  Decision-Making and Rule based learning
Probe Tasks | Administered pre testing, at 2 weeks, 3 weeks and after completion of training at 6 weeks
  Decision-Making and Rule based learning
WHO BREF Quality of Life | before and after training, at 6 weeks
  general quality of life
Dysexecutive Questionnaire | pre and post training, at 6 weeks
  Test of everyday executive functioning behaviors; self and informant reports

OTHER OUTCOMES:
Cognitron Cognitive Assessment Battery | Pre & Post Testing, after completion of training at 6 weeks
  Tests of memory, reaction time, and executive Functioning
fNIRS | pre and post training testing, after completion of training at 6 weeks
  Functional spectroscopy of oxygenated and deoxygenated hemodynamic responses

CONTACTS AND LOCATIONS:
Overall Officials: Fofi Constantinidou, Ph.D., Principal Investigator — University of Cyprus
Locations (1):
- University of Cyprus, Nicosia, Cyprus, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be entered in an open access depository as per funding agency's requirements. IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: After data has been published, December 2026.
Access Criteria: upon request
URL: https://www.ucy.ac.cy/brainn/

REFERENCES:
- See also: Project website — http://ucy.ac.cy/brainn